CLINICAL TRIAL: NCT05651308
Title: Improving How People Living With Dementia Are Selected for Care Coordination: A Pragmatic Clinical Trial Embedded in an Accountable Care Organization
Brief Title: Improving How People Living With Dementia Are Selected for Care Coordination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-10025292; 3U54AG063546-03 (NIH); Subaward 00002102 (Other Grant/Funding Number: Brown University)
Record Dates: First submitted 2022-12-05; First posted 2022-12-15 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Dementia
Keywords: care coordination; accountable care organization
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will assign care coordinators to PLWD based on perceived need for assistance with care coordination. Perceived need will be measured through a proxy's responses to a previously validated telephone survey on perceptions of care coordination.
  Interventions: Behavioral: Care coordination delivered based on perceived need
- Control (Active Comparator): Usual care assigns patients to care coordinators in response to a discharge from a hospital or a direct referral from a physician.
  Interventions: Behavioral: Care coordination delivered based on usual care (e.g. discharge from hospital)

INTERVENTIONS:
Behavioral: Care coordination delivered based on perceived need — If proxies for patients in intervention group report on the survey that they experience difficulty coordinating care among the patients' providers, the patient will be selected for care management services. Those services will attempt to address the problems with care coordination that the proxy reported.
  Arms: Intervention
Behavioral: Care coordination delivered based on usual care (e.g. discharge from hospital) — If a patient is discharged from a hospital, the patient will be selected for care management services.
  Arms: Control

SUMMARY:
Many people living with dementia (PLWD) and their care partners may benefit from the assistance of a care coordinator, a member of the medical team who facilitates communication among all the people involved. However, care coordinators' time is limited, and there is uncertainty about which patients should be selected to receive their help. This pragmatic clinical trial embedded in an accountable care organization will determine the comparative effectiveness of two approaches for assigning care coordinators to PLWD.

DETAILED DESCRIPTION:
This project will use a pragmatic clinical trial embedded in an accountable care organization (ACO) to determine the comparative effectiveness of two different approaches for selecting PLWD to receive support from care coordinators: (1) an approach that assigns PLWD to care coordinators based on care partners' self-reported difficulty with care coordination, or (2) usual care, which generally assigns PLWD to care coordinators after hospital discharge, regardless of perceived need. The investigators will include community-dwelling Medicare beneficiaries ≥65 years old with dementia who have been attributed to the NewYork Quality Care ACO and who have fragmented care. The investigators will randomize the participants into two groups. This study is highly pragmatic, and the intervention is sustainable and scalable. Moreover, the proposed approach has the potential to improve care delivery and outcomes for PLWD.

ELIGIBILITY:
Inclusion Criteria:

* Medicare beneficiaries ≥65 years old who:
* Are attributed to the NewYork Quality Care accountable care organization by Medicare,
* Have dementia (as measured in claims using the Bynum standard 1-year definition),
* Reside in the community, and
* Had fragmented ambulatory care in the previous 12 months (defined as a reversed Bice-Boxerman Index greater than or equal to the median score for this population, using Medicare claims)

Exclusion Criteria:

* Those who reside in long-term care or nursing home facilities (based on addresses in Medicare claims), or
* Enrolled in home hospice

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 385 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Kern, MD, MPH, Principal Investigator — Weill Medical College of Cornell University; Vincent Mor, PhD, Study Director — Brown University
Locations (1):
- New York Presbyterian Hospital - Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 193 | 192
Completed | 193 | 192
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 193 | 192 | 385
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.8 (6.9) | 82.3 (7.0) | 82.6 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 108 | 217
  Male | 84 | 84 | 168
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 154 | 153 | 307
  Non-White | 39 | 39 | 78
Medicare enrollment type [Count of Participants; unit: Participants]
  Aged duals | 48 | 33 | 81
  Aged non-duals | 141 | 158 | 299
  End-stage renal disease | 4 | 1 | 5
  Disabled | 0 | 0 | 0
Co-morbidities [Count of Participants; unit: Participants]
  Acute myocardial infarction | 10 | 7 | 17
  Atrial fibrillation | 32 | 18 | 50
  Chronic kidney disease (any stage other than ESRD) | 50 | 51 | 101
  Chronic obstructive pulmonary disease or bronchiectasis | 28 | 28 | 56
  Colorectal cancer | 15 | 6 | 21
  Depression | 65 | 57 | 122
  Diabetes | 39 | 38 | 77
  Endometrial cancer | 4 | 3 | 7
  End-stage renal disease (ESRD) | 3 | 3 | 6
  Female or male breast cancer | 18 | 15 | 33
  Heart failure | 63 | 51 | 114
  Hyperlipidemia | 123 | 123 | 246
  Hypertension | 130 | 122 | 252
  Ischemic heart disease | 86 | 81 | 167
  Lung cancer | 6 | 2 | 8
  Prostate cancer | 13 | 17 | 30
  Stroke / transient ischemic attack | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Emergency Department Visits or Hospital Admissions
Description: Occurrence of an emergency department visit or hospital admission, as measured in Medicare claims
Time Frame: Over 12 months (beginning 1 month after the start of care coordination)
Population: Intention-to-treat analysis
Measure: Number (95% Confidence Interval); unit: events per 100 person-days alive
Arm/Group | Intervention | Control
Number analyzed (Participants) | 193 | 192
events per 100 person-days alive | 0.33 [0.28 to 0.39] | 0.35 [0.30 to 0.41]

2. Secondary Outcome: Acceptability
Description: The number of people who accepted care management in each group
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 193 | 192
Participants | 19 | 14
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.37, Chi-squared; Risk Difference (RD) = 0.026, 95% CI 2-sided [-0.03 to 0.08] — Risk difference = Intervention proportion minus control proportion

3. Secondary Outcome: Appropriateness
Description: The number of people with problems in scope for care coordinators, out of all people who received care management
Time Frame: Up to 1 year
Population: The only participants who were analyzed in this measure were those who received care management services (as shown in Secondary Outcome #1).
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 14
Participants | 19 | 14

4. Secondary Outcome: Fidelity
Description: The number of people who actually received care coordination services, out of all of those who agreed to receive it
Time Frame: Up to 1 year
Population: The only people analyzed for this measure were people who agreed to receive care management (as shown in Secondary Outcome #1).
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 14
Participants | 19 | 14

5. Secondary Outcome: Efficiency
Description: The number of care coordinator encounters in each group. This measure allows more than one encounter per person.
Time Frame: Up to 1 year
Measure: Number; unit: Encounters
Arm/Group | Intervention | Control
Number analyzed (Participants) | 193 | 192
Encounters | 77 | 54

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 32/193 | 37/192
Serious Adverse Events (participants affected / at risk) | 52/193 | 45/192
Other Adverse Events (participants affected / at risk) | 47/193 | 57/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=193) | Control (N=192)
All-cause hospitalization (General disorders) | 52 (90) | 45 (74)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=193) | Control (N=192)
Emergency department visit (General disorders) | 47 (63) | 57 (84)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT05651308/Prot_SAP_000.pdf